CLINICAL TRIAL: NCT00710645
Title: Assessment of Spasticity in MS Patients Using a Lido Workset
Brief Title: Lido Workset Study
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200310977
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Spasticity
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm I: 50 subjects with multiple sclerosis will be tested one time on the Lido Workset. The test will take approximately 25 minutes. The servo-controlled torque motor system will analyze resistance to passive movement of the knee. This testing may be repeated for a group of randomly selected subjects. Each subject will be given the option to participate in the extended testing or to decline. The testing for this subset of subjects will be done as follows: first session, second session one week after the first session, third session three weeks after the first session. The total length of time for participation in this study may be up to three weeks.
  Interventions: Device: Lido Workset
- Arm II: 25 normal subjects will be tested on the Lido workset. The testing will be performed one time for each patient and will take approximately 25 minutes. The servo-controlled torque motor system will analyze resistance to passive movement of the knee. This testing may be repeated for a group of randomly selected control subjects. Each subject will be given the option to participate in the extended testing or to decline. The testing for this subset of subjects will be done as follows: first session, second session one week after the first session, third session three weeks after the first session. The total length of time for participation in this study may be up to three weeks.
  Interventions: Device: Lido Workset

INTERVENTIONS:
Device: Lido Workset — The intervention will consist of spasticity testing on the Lido Workset device. The servo-controlled torque motor system will analyze resistance to passive movement of the knee.

SUMMARY:
This is a single-site, pilot study. In this study, we hope to learn if the Lido Workset is a sensitive measure of limb spasticity in patients with Multiple Sclerosis (MS). The Lido Workset is a FDA approved, non-invasive device which has been used to assess motor function and spasticity. The testing will take approximately 25 minutes. Subjects will lie down on a table and have a leg attached to the Lido Workset device arm. The Lido Workset will move the leg back and forth many times at different speeds. The Lido Workset will also analyze resistance to passive (while subject is not moving or resisting movement) movement of the wrist and knee.

DETAILED DESCRIPTION:
The information gathered from testing individuals with spasticity due to multiple sclerosis with the Lido Workset has been important in making adjustments to the Lido Workset to show a greater degree of sensitivity in assessing varying degrees of spasticity.

Healthy control subjects will be used to compare the spasticity data of multiple sclerosis subjects with subjects with normal muscle tone to determine the sensitivity of the Lido measurements.

The testing will be performed one time for each patient and will take approximately 25 minutes. The servo-controlled torque motor system will analyze resistance to passive movement of the knee. This testing may be repeated for a group of randomly selected subjects from both the MS subjects and control subjects. The testing for this subset of subjects will be done as follows: first session, second session one week after the first session, third session three weeks after the first session. The total length of time for participation in this study may be up to three weeks. This additional testing will be done in order to compare the results with the Lido data obtained at similar timepoints from the subjects enrolled in the Cannabis for Spasticity in MS study. Each subject will be given the option to participate in the extended testing or to decline.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of multiple sclerosis and
* Must have some degree of spasticity or
* Must be a healthy control subject
* Ability to give informed consent

Exclusion Criteria:

* Patients with any life-threatening or unstable clinically significant disease
* Patients with other causes of reduced range of motion of the knee or wrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be men and women diagnosed with Multiple Sclerosis who have some degree of spasticity in the knee or wrist. They must be at least 18 years of age. This study will also enroll healthy controls who are able to give consent and who are at least 18 years of age. Subjects will be recruited from the community and from the PI's clinic population.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2003-04; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Assess measure of spasticity | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Agius, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No